CLINICAL TRIAL: NCT00598117
Title: Quality Of Life Outcomes Following Treatment for Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-083
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer
Keywords: Esophageal; CancerEsophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Group 1 (newly diagnosed patients) Initial assessment → first post op visit → 6 and 12 months post surgery
  Interventions: Behavioral: Questionnaires
- 2: Group 2 (post-treatment patients) A one-time assessment will be conducted at least 18 months following treatment
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Newly diagnosed patients will be assessed at four points Time 1 (prior to treatment)
  * Initial QOL form
  * FACT-E, PAR, Symptom Assessment Scale, MDSS, Time 2 (initial post-op)
  * Follow up QOL form
  * FACT-E, PAR, Symptom Assessment Scale, MDSS Time 3 (6 months post op)
  * Follow up QOL form
  * FACT-E, PAR, Symptom Assessment Scale, MDSS, Time 4 (1 year post op)
  * Follow up QOL form
  * FACT-E, PAR, Symptom Assessment Scale, MDSS

SUMMARY:
The goal of this study is to evaluate how treatment for esophageal cancer affects your quality of life. The findings of this study may help us understand how this disease and its treatment affect your lifestyle, diet, exercise, support system and overall quality of life. We hope this study will provide important information that can be used to develop programs to improve the quality of life of patients with esophageal cancer.

DETAILED DESCRIPTION:
In order to determine the impact of esophageal cancer and its treatment on patients' quality of life over time, this study will prospectively follow a cohort of patients at specified intervals, evaluating their physical symptoms, physical and social functioning and overall quality of life. Medical and sociodemographic factors as well as health behaviors that might be predictive of adaptation will be tested. This is a preliminary investigation and it is hoped that we will be able to base future research questions on the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of esophageal cancer.
* Anticipated to undergo surgical resection (Ivor Lewis, Trans Hiatal, McKeown procedure) of esophageal cancer. (Group 1 patients only)
* Underwent esophagectomy for esophageal cancer at least 18 months prior to consent, with no evidence of disease. (Group 2 patients only)
* Ability to speak, read and write English.

Exclusion Criteria:

* Inability to give informed consent.
* Patients anticipated to require a laryngectomy as part of their surgical resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a descriptive study comprising two cohorts of esophageal cancer patients. The first cohort will be followed prospectively and will include patients newly diagnosed with esophageal cancer prior to treatment. QOL assessments will be administered pre-surgery, at first post-operative visit, and at 6 and 12 months post surgery. The second cohort will be a cross sectional sample and include patients more than 18 months post treatment, without evidence of disease who will undergo one QOL assessment. This is a preliminary investigation and it is hoped that we will be able to base future research questions on our results of this study.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2003-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To prospectively evaluate the quality of life of patients before and after esophageal cancer resection. | Initial assessment → first post op visit → 6 and 12 months post surgery

SECONDARY OUTCOMES:
To describe a cohort of long term survivors of esophageal cancer in order to identify significant features in patients more than 18 months post surgery. | 18 months following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Manjit Bains, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org